CLINICAL TRIAL: NCT04397731
Title: Role of Endoscopic Ultrasound-guided Fine-needle Biopsy in the Diagnosis of Autoimmune Pancreatitis
Brief Title: Prospective Study on the Role of Eus-fnb in the Diagnosis of Autoimmune Pancreatitis
Acronym: BIO_AIP
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Stefano Francesco Crinò, MD, MD, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 2482CESC
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2021-03

CONDITIONS: Autoimmune Pancreatitis
Keywords: ICDC criteria; AIP; HISTOLOGY IN AIP; EUS-FNB; Endoscopic fine needle biopsy
MeSH Terms: conditions — Autoimmune Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the reported histological procurement yield of the end-cutting needles, the investigators supposed that the use of EUS-FNB in probable AIP patients, generally aimed only to rule-out malignancy, could provide histological tissue samples useful in enhancing the diagnostic level reached without histology, or defining the type of AIP.

DETAILED DESCRIPTION:
The primary aim is to evaluate the capability of EUS-FNB to enhance diagnostic levels of AIP, that means to obtain definitive diagnosis of type 1 and type 2 AIP. Secondary aims are to evaluate: Safety of EUS-FNB in this setting of patients; the possibility to obtain a definitive diagnosis in focal/segmental form of AIP (that are the most clinically relevant because of the mimicking of cancer); diagnostic yield of EUS-FNB in this patient population; the rate of pancreatic neoplasms mimicking AIP.

Consecutive patients ≥ 18 years old, with suspected focal or diffuse AIP, according to ICDC (probable type 1 AIP; probable type 2 AIP; NOS-AIP) with written consent to participate in the study will be enrolled.

Exclusion criteria include: previous diagnosis of AIP; definitive type 1 AIP; steroid administration within 3 months before the EUS-FNB; coagulation disorders; pregnancy and lactation; unability to give informed consent .

The histopathology of the preparations will be evaluated, according to the ICDC, including the LPSP findings and the IDCP findings and recording the absence or presence of specific criteria: Periductal lymphoplasmacytic infiltrate without GELs, Storiform fibrosis, Obliterative phlebitis >10 IgG4-positive cells per HPF; GEL of duct wall; Granulocytic and lympho- plasmacytic acinar infiltrate.

According to the current clinical practice, when the diagnosis of AIP is confirmed (and malignancy is ruled-out) patient will be treated with the standard therapy for AIP. Patients will be followed for 12 months, in order to exclude misdiagnosed malignancy, and to evaluate the clinical course of the disease (response to steroid therapy, relapses, changes in imaging findings or surgical pathology in resected patients).

The final diagnosis of AIP will be confirmed on surgical pathology (in resected patients) or when a compatible clinical course is observed during a follow-up of at least 1 year (significant improvement on imaging after steroid therapy, no appearance of metastasis or sign of infiltration).

The number of cases where EUS-FNB histology improves the diagnostic level will be summarized using absolute and relative frequencies. The 95% confidence interval of this proportion will also be computed. The number of adverse events, the number of cases where histological finding diagnostic of AIP are observed in focal/segmental form and the number of pancreatic neoplasm will be summarized using absolute and relative frequencies. Sensitivity, specificity, positive likelihood ratio (LR+), negative likelihood Ratio (LR-) and the ROC curve will be used to analyze the capability of EUS-FNB to obtain a definitive diagnosis of type 1 and 2 AIP.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients ≥ 18 years old;
* Suspected focal or diffuse AIP, according to ICDC:

Probable type 1 AIP Probable type 2 AIP NOS-AIP

• provision of written consent to participate in the study.

Exclusion Criteria:

* Previous diagnosis of AIP
* Definitive type 1 AIP
* Steroid administration within 3 months before the EUS-FNB
* Coagulation disorders
* Pregnant and lactating women
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected AIP who need histological sampling for diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The primary aim is to evaluate the capability of EUS-FNB to enhance diagnostic levels of AIP, that means to obtain definitive diagnosis of type 1 and type 2 AIP. | 2 years
  For the primary aim, the endpoint is the percentage of cases where EUS-FNB histology improve the diagnostic level:
  * from a probable AIP 1 to definitive AIP 1 (i.e., percentage of type 1 Level 1 H);
  * from a probable AIP 2 to definitive AIP 2 (i.e., percentage of type 2 Level 1 H);
  * from an AIP-NOS to AIP 1 or 2 (i.e., percentage of type 1 and 2, Level 1 H or Level 2 H).

SECONDARY OUTCOMES:
Safety of EUS-FNB in AIP patients: percentage of adverse events observed | 2 years
  The percentage of adverse events observed
The possibility to obtain a definitive diagnosis in focal/segmental form of AIP (that are the most clinically relevant because of the mimicking of cancer). | 2 years
  The Percentage of cases where histological finding diagnostic of AIP (Level 1 and Level 2) are observed in focal/segmental form.
Diagnostic yield of EUS-FNB in this patient population. | 2 years
  The sensitivity, specificity, PPV, NPV, and accuracy calculated in comparison with the final diagnosis
The rate of pancreatic neoplasms mimicking AIP | 2 years
  The percentage of pancreatic neoplasm in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Francesco Crinò, Principal Investigator — Azienda Ospedaliera Integrata Verona
Locations (2):
- Azienda Ospedaliera Integrata Verona, Verona, Italy
- Tsukasa Ikeura, Osaka, Japan

REFERENCES:
- [Derived] Conti Bellocchi MC, Crino SF, Ikeura T, Carrara S, Oh D, Nakamaru K, Terrin M, Song TJ, Caldart F, Sina S, De Pretis N, Manfrin E, Frulloni L. Impact of EUS-guided fine-needle biopsy sampling on International Consensus Diagnostic Criteria for diagnosing autoimmune pancreatitis: a prospective multicenter study. Gastrointest Endosc. 2025 Oct;102(4):559-568.e1. doi: 10.1016/j.gie.2025.02.038. Epub 2025 Feb 28. PMID 40024297